CLINICAL TRIAL: NCT00224198
Title: Evaluation of the Lungs of Individuals With Lung Disease With Segmental Bronchopulmonary Lung Lavage, Bronchial Brushing and Bronchial Wall Biopsy
Brief Title: Evaluation of the Lungs of Individuals With Lung Disease
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 0005004440
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-04

CONDITIONS: Lung Disease; Bronchitis; Emphysema; COPD; Asthma
MeSH Terms: conditions — Lung Diseases; Bronchitis; Emphysema; Pulmonary Disease, Chronic Obstructive; Asthma | interventions — Bronchoscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Specimens will be retained from both a blood draw and a bronchoscopy procedure.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Lung Disease: All study individuals will be males or females that are 18 years or older and are able to provide informed consent and have been diagnosed with lung disease.
  Interventions: Procedure: Lung Disease

INTERVENTIONS:
Procedure: Lung Disease — Bronchoscopy consists of the passage via the mouth or nose of a flexible fiberoptic bronchoscopy into the airways. In the lavage (washing) procedure, sterile 0.9% saline (5 x 20 ml aliquots in 1 to 3 sites) is instilled into the lung and immediately suctioned back, washing off cells lining the airways.In the brushing procedure, a small cytology brush is passed through the bronchoscope, and a small area of the airway wall is brushed gently to obtain epithelial cells lining the airway. Certain individuals may have bronchial wall biopsy carried out. In this procedure, a small biopsy forceps is passed through the bronchoscope and a small biopsy is obtained from the bronchial wall.
  Other Names: Bronchoscopy

SUMMARY:
The purpose of this protocol is to obtain biologic materials from the blood and lungs from patients with lung disease in order to develop an understanding of the etiology and pathogenesis of these disorders. General admission criteria for this project will require at least one of the following: (1) symptoms consistent with pulmonary disease; (2) chest X-ray consistent with lung disease; (3) pulmonary function tests consistent with lung disease; (4) lung biopsy consistent with lung disease; (5) family history of lung disease; and (6) patients with diseases of organs with known association with lung disease.

DETAILED DESCRIPTION:
Patients will undergo a general medical evaluation by a pulmonary physician (and consultants as appropriate for other organs). The typical routine medical studies to be carried out may include: chest X-ray (posterior-anterior and lateral), non-contrast high resolution CT scan of the chest, pulmonary function tests, electrocardiogram, echocardiogram, general hematologic studies, general serologic studies, /immunologic studies, biochemical analyses (including carboxyhemoglobin to measure blood carbon monoxide levels in order to accurately evaluate the diffusion capacity in individuals who smoke since smoking increases the blood levels of carbon monoxide), alcohol blood test, urinalysis, urine chemistries (including blood or urine nicotine and cotinine test to evaluate urine for active or passive exposure to nicotine), blood or urine drug screening (to evaluate use of recreational drugs and/or mood altering medications), pregnancy test (if applicable) and HIV serology. Also, a sweat chloride and sweat rate test may be performed by the physician to evaluate participants with a possible diagnosis of cystic fibrosis.

The study individual will undergo fiberoptic bronchoscopy with a combination of bronchial brushing and/or bronchoalveolar lavage and/or bronchial wall biopsy. The primary factor for determining if an individual will have bronchial alveolar lavages (BAL) and/or brushings and/or biopsies is the particular lung disease affecting the individual. This will depend on the known mechanism relevant to the pathogenesis of the particular disease. For example, in individuals with asthma, the samples may include airway brushing and airway biopsies; in contrast, in individuals with chronic obstructive pulmonary disease (COPD), sampling may include airway brushings, airway biopsies, and bronchoalveolar lavage. Other determining factors include: the amount of moderate sedation (if used) and the amount of analgesia used; the maximal dosage of topical lidocaine that is allowed per procedure; allergic reactions to any of the medications used in the procedures; and individual's tolerance to the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Must provide informed consent
* Males and females, age 18 years and older
* Lung disease proven by at least one of the following: (1) symptoms consistent with pulmonary disease; (2) chest X-rays consistent with lung disease; (3) pulmonary function tests consistent with lung disease; (4) lung biopsy consistent with lung disease; (5) family history of lung disease; and (6) diseases of organs with known association with lung disease
* Must provide HIV informed consent

Exclusion Criteria:

* Any history of allergies to xylocaine, lidocaine, versed, valium, atropine, pilocarpine, isoproterenol, terbutaline, aminophylline, or any local anesthetic will not be included in the study
* Drug and/or alcohol abuse within the past six months
* Females who are pregnant or nursing
* Individuals who test positive for HIV (other than for studies directly related to the HIV virus)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The source of potential subjects will be the population of individuals defined by the eligibility criteria below, individuals in the New York metropolitan area and elsewhere. Up to one hundred volunteers will take part in the study each year. Accrual will be random with no bias as to gender or racial/ethnic group. All study individuals will be males or females that are 18 years or older and are able to provide informed consent. Advertisements will be posted at various educational institutions and hospitals and placed in newspapers in the New York metropolitan area. Paid volunteer referrals will also be used for patient recruitment.
Sampling Method: Non-Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2004-01; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Understand lung disease etiology and pathogenesis | 9/31/2012
  The primary objective is to develop and understand the etiology and pathogenesis of these lung disease disorders.

SECONDARY OUTCOMES:
Identify suitable candidates | 9/31/2012
  The secondary objective is to identify individuals who will be suitable candidates for other protocols such as those involving investigational new drugs.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G Crystal, MD, Principal Investigator — Department of Genetic Medicine, WMC of Cornell University
Locations (1):
- Department of Genetic Medicine, Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang G, Wang R, Ferris B, Salit J, Strulovici-Barel Y, Hackett NR, Crystal RG. Smoking-mediated up-regulation of GAD67 expression in the human airway epithelium. Respir Res. 2010 Oct 29;11(1):150. doi: 10.1186/1465-9921-11-150. PMID 21034448
- [Derived] Carolan BJ, Harvey BG, Hackett NR, O'Connor TP, Cassano PA, Crystal RG. Disparate oxidant gene expression of airway epithelium compared to alveolar macrophages in smokers. Respir Res. 2009 Nov 17;10(1):111. doi: 10.1186/1465-9921-10-111. PMID 19919714